CLINICAL TRIAL: NCT02788630
Title: Infant Sleep Hygiene Counseling: A Randomized Controlled Trial
Brief Title: Infant Sleep Hygiene Counseling Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Collaborators: University of Toronto (Other); University of Sao Paulo (Other); Hospital Nossa Senhora da Conceicao (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Iná da Silva dos Santos, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 47/2014
Record Dates: First submitted 2016-05-18; First posted 2016-06-02 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Arm: Experimental: Intervention group Field workers trained in sleep hygiene counseling will advice the mothers randomly allocated to the intervention group. The intervention will be delivered at the child household and will include information on: Normal sleep behaviors during the first year of life; ideal conditions to promote sleep onset like environmental improvements that ensure restful sleep (no screen media, low noise and light); calming naptime routines and avoiding stimulating or stressing children just before naptime; practices that promote child self-regulation of sleep, including putting infants to sleep drowsy but awake; and how to handle nighttime awakenings. A booklet with the intervention content to aid the mother in implementing the intervention will be used.
  Interventions: Behavioral: Sleep hygiene counseling
- Control group (No Intervention): Mothers randomly allocated to the control group will be visited at home following the same schedule as the intervention group. The control group will receive a written material describing the advantages of breastfeeding over maternal and child health. No advice in relation to child sleep hygiene will be delivered to the mothers from the control group.

INTERVENTIONS:
Behavioral: Sleep hygiene counseling — The mothers of the eligible infants will be visited at home and will be invited to participate at the study. To those who sign the Consent Form (CF) a following visit will be scheduled to within 5 days. Between CF signature and the 5-day visit, the enrolled children will use an actigraph-device in the leg and the mothers will fill out a sleep diary registering the times of the day the child is asleep, awake, napping, and feeding. At the 5-day visit the child allocation in the trial (intervention or control group) will be uncovered and the sleep recommendations will be delivered to mothers in the intervention group. Phone calls on days 6 and 7 and a home visit on day 8 will be paid to support mothers for possible difficulties in implementing the recommendations.
  Other Names: Child sleep trial
  Arms: Intervention group

SUMMARY:
This study will evaluate the efficacy of an intervention to improve quality and duration of self-regulated nighttime sleep (the amount of time the child maintains a combination of uninterrupted sleep, quiet wakefulness, and re-initiation of sleep without parental intervention).

DETAILED DESCRIPTION:
The development of adequate sleep patterns is paramount to the optimal neurodevelopment, as well as to promote proper learning, develop memory and preserve cerebral plasticity. Factors that hinder sleep patterns can negatively influence the child's growth, neurological and motor development.

The investigators will conduct a randomized controlled trial within the 2015 Pelotas Birth Cohort. At the 3-month follow-up, children who sleep less than 13 hours per 24 hours (nighttime sleep and daytime naps) will be eligible for the study. The sample size was estimated at 276 children per arm. Nighttime self-regulated sleep duration will be evaluated at baseline (age 3 months) and at 6, 12 and 24 months using actigraphy and via a sleep diary completed by the mother. Following block randomization, mothers from the intervention group will be visited by a trained fieldworker who will deliver counseling on age-appropriate normal sleep behaviors, how to facilitate sleep onset and how to manage night awakenings.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to the trial the child will need to belong to the Pelotas 2015 Birth Cohort, to be born healthy (newborns that needed intensive care after birth and with any congenital malformations will be excluded) from a single pregnancy at gestational age 37 weeks or greater, and to sleep regularly on average less than 13 hours per 24 hours (daytime and nighttime sleep) at three months of age (as reported by the mother). The information on child sleep duration per 24 hours will be gathered during the interview with mothers from the entire cohort, by means of the answer to the questions: "How many hours does the child sleep from 7pm to 7am?" and "How many hours does the child sleep from 7am to 7pm?"as well as number and duration of daytime naps, number of wake episodes during the night and how long it takes to the child to fall sleep after a nocturnal awakening.

Exclusion Criteria:

* Because the potential effect of the programmed maternal physical activity during pregnancy over the sleep duration or over the poor-sleeper-newborn answer to the sleep trial is not known, newborns to mothers that participated at the PAMELA trial will not be eligible to the sleep trial. The PAMELA (Physical Activity for Mothers Enrolled in Longitudinal Analysis) is a randomized controlled trial nested in the Pelotas 2015 birth cohort planned to assess the effect of regular exercise during pregnancy on the prevention of hypertension, pre-eclampsia and preterm birth. Eligible pregnant women between the 16th and 20th week of gestation are allocated into control group (426 women who are advised to keep their usual daily activities) or intervention group (213 women who engage in an exercise program, three sessions a week).

Also, because the sleep intervention will recommend a series of environmental improvements to ensure a restful sleep (no screen media, low noise and light), the intervention will be restricted to families living in households with at least one bedroom. Children in continued use of medicines that can alter the sleep architecture and/or lead to drowsiness, like anticonvulsivants, will be excluded.

Ages: 3 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Nighttime self-regulated sleep duration at 6, 12 and 24 months of age | Up to 24 months
  Nighttime self-regulated sleep duration is the maximum amount of time the child stays asleep or awake without awakening the parents at ages 6, 12 and 24 months. This outcome will be evaluated by using the actigraphy and diary records for 5 days. The Brief Infant Sleep Questionnaire (BISQ) will be used at these three visits.

SECONDARY OUTCOMES:
Linear growth between age 3-12 and 12-24 months of age | Up to 24 months
  The effect of the intervention on linear growth will be estimated by comparing conditional growth between groups. At 3, 12 and 24 months of age anthropometric evaluation will include measures of length and weight. Length will be measured using a foldable wooden infantometer, custom made for the study, using for measurement a nylon tape measure with 1 mm precision adhered to a groove carved into the body of the instrument. Mother and child weight will be measured using an electronic scale (150 kg capacity and 100 g precision), the mother being weighed first alone then holding the baby. The child's weight will be calculated as the difference between the two measures. The mother will be weighed clothed, but without heavy outfits, and clothes worn by the mother will be recorded. The child will be weighed undressed, whenever allowed by the mother. Otherwise, the child's clothing will be recorded.
Neurocognitive development at 12 and 24 months of age. | Up to 24 months
  The holistic neurodevelopment assessment designed and implemented by the Intergrowth-21st Project (Intergrowth neurodevelopment assessment tool - INTER-NDA) will be used to measure cognitive, motor, language, behavioral, attention, and executive function outcomes in children at 24 months. The recently developed 12-month version of the instrument (Oxford neurodevelopment assessment tool - OX-NDA) will be used to assess the child neurodevelopment at 12 months of age.
Validation study of the Oxford neurodevelopment assessment tool (OX-NDA) | Up to 12 months
  100 children aged 10-12 months from the 2015 Pelotas Birth Cohort will participate in a validation study in which the OX-NDA results will be compared to the results of the Bayley Scales of Infant and Toddler Development - Third Edition (BSDI-III) taken as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Del Ponte, PhD, Study Chair — Federal University of Pelotas; Suélen Cruz, PhD, Study Chair — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Santos IS, Del-Ponte B, Tovo-Rodrigues L, Halal CS, Matijasevich A, Cruz S, Anselmi L, Silveira MF, Hallal PRC, Bassani DG. Effect of Parental Counseling on Infants' Healthy Sleep Habits in Brazil: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1918062. doi: 10.1001/jamanetworkopen.2019.18062. PMID 31860110
- [Derived] Santos IS, Bassani DG, Matijasevich A, Halal CS, Del-Ponte B, da Cruz SH, Anselmi L, Albernaz E, Fernandes M, Tovo-Rodrigues L, Silveira MF, Hallal PC. Infant sleep hygiene counseling (sleep trial): protocol of a randomized controlled trial. BMC Psychiatry. 2016 Sep 2;16(1):307. doi: 10.1186/s12888-016-1016-1. PMID 27590170